CLINICAL TRIAL: NCT01405625
Title: Improving Parent Understanding of Instructions About Asthma Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 09-0358
Record Dates: First submitted 2011-07-26; First posted 2011-07-29 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: Asthma; Health literacy; Parent knowledge of appropriate action plan steps
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAAAI Action Plan (Active Comparator): Asthma Action Plan from the American Academy of Allergy, Asthma, and Immunology
  Interventions: Other: AAAAI standard of care written action plan
- Asthma pictogram written action plan (Experimental): Cartoon/pictogram-based written action plan sheet
  Interventions: Other: Pictogram-based asthma action plan

INTERVENTIONS:
Other: Pictogram-based asthma action plan — Asthma action plan using plain language, pictograms, and photographs
  Arms: Asthma pictogram written action plan
Other: AAAAI standard of care written action plan
  Arms: AAAAI Action Plan

SUMMARY:
Asthma has an especially great impact on poor urban children and their families. In addition to higher asthma prevalence and morbidity, those in low SES urban areas are at risk for low health literacy. Low health literacy is associated with poorer asthma outcomes. The provision of a written asthma action plan has been shown to help with asthma management and to reduce hospitalizations and ER visits. Poor urban families who may have low literacy may need an alternative asthma action plan to convey the treatment plan.

This pilot study proposes to investigate whether a plain language asthma action plan can improve parent understanding and adherence with medication instructions, compared to standard written materials, among parents of children with asthma. This is an RCT in which parents of children with asthma will be randomized to either receive a pictogram-based low literacy asthma action plan, or a standard action plan (AAAAI), to examine whether those who receive the low literacy plan have improved asthma action plan knowledge when presented with a hypothetical scenario.

A second part of the study is to examine whether providers who are given the pictogram-based low literacy asthma action plan will be more likely to counsel about certain aspects of asthma management (eg. need for daily medications even when sick, spacer use, confusion between everyday and rescue inhaler)compared to providers who receive use a standard action plan (AAAAI). This is an RCT in which pediatric providers are randomized to counsel a hypothetical patient using the pictogram-based action plan or the standard action plan (AAAAI).

ELIGIBILITY:
Parent study:

Inclusion Criteria:

* Primary caregiver / parent / legal guardian of child 2-12 years old
* Child with diagnosis of asthma

Exclusion Criteria:

* Parent not English or Spanish-speaking

Provider study:

Inclusion Criteria:

* Health providers who care for children with asthma

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Asthma Action Plan knowledge (parent) | 1 day (on same day of enrollment; no outcome assessment after day of enrollment)
  Outcome measure will be assessed on the day of enrollment only, using a hypothetical scenario. No outcome assessments will be performed after the day of enrollment.

SECONDARY OUTCOMES:
Asthma action plan content (provider) | same day as presentation of hypothetical counseling scenario
  Provider coverage of green/yellow/red zone concepts, spacer use, medication information, symptoms; use of low literacy principles

CONTACTS AND LOCATIONS:
Overall Officials: Suzy Tomopoulos, MD, Principal Investigator — NYU School of Medicine; Shonna (Hsiang) Yin, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States